CLINICAL TRIAL: NCT03318887
Title: Sofosbuvir Plus Daclatasvir With or Without Ribavirin for Chronic Hepatitis C Infection: Impact of Drug Concentration on Viral Load Decay
Brief Title: Impact of Sofosbuvir and Daclatasvir Concentration on HCV RNA
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2016_001
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
Keywords: Cirrhosis; Direct acting antiviral agents; Hepatitis C; Pharmacological monitoring
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Sofosbuvir; daclatasvir; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sofosbuvir/daclatasvir: Patients with hepatitis C virus (HCV) infection treated with sofosbuvir/daclatasvir combination therapy with or without ribavirin between February and September 2014
  Interventions: Drug: Sofosbuvir/daclatasvir with or without ribavirin

INTERVENTIONS:
Drug: Sofosbuvir/daclatasvir with or without ribavirin — Direct-acting antiviral treatment for hepatitis C virus infection
  Other Names: Combination of sofosbuvir and daclatasvir with or without ribavirin

SUMMARY:
Sofosbuvir plus daclatasvir with or without ribavirin is one of the currently recommended treatment option for chronic hepatitis C. The objectives were to identify factors associated with sofosbuvir/daclatasvir plasma concentrations variations and to evaluate their impact on viral kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatitis C virus infection treated with sofosbuvir/daclatasvir
* Patients with at least one measurement of sofosbuvir or daclatasvir plasma concentration
* Follow-up of at least 3 months after the end of treatment

Exclusion Criteria:

* Patients with severe renal failure (estimated glomerular filtration rate (eGFR)<30ml/min/1.73m2)
* Patients with liver transplantation during therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HCV infected patients from the Department of Hepatology, Croix-Rousse Hospital, Lyon, France receiving sofosbuvir/daclatasvir with or without ribavirin between February and September 2014 were considered
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Sofosbuvir/daclatasvir plasma concentration | Sofosbuvir/daclatasvir plasma concentrations were measured at week 4, 8, 12 and 24 during therapy

SECONDARY OUTCOMES:
HCV viral load | At treatment initiation, at week 4, 8, 12 and 24 of therapy and 12 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Zoulim, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No